CLINICAL TRIAL: NCT03619447
Title: Comparison of the Ultrasound Guided Erector Spinae Plane Block Versus Serratus Plane Block in Totally Mastectomy
Brief Title: Comparison of ESP Block Versus Serratus Block
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, ebru biricik, Anesthesiologist, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESP vs Serratus
Record Dates: First submitted 2018-08-02; First posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Both participants and anaesthesia provider will not know which intervention applied. Another anaesthesia provider who did not perform any block will follow and record to the study data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESP block group (Active Comparator): Under general anaesthesia, Ultrasound guided ESP block will perform at the T6 level with15 ml bupivacain+ 5ml lidocaine, bilaterally. Morphine 0.1 mg/kg will administer at last 30 minutes of surgery for postoperative analgesia. Patient controlled analgesia (PCA) with morphine will apply to the all patients. Postoperative pain assessment and morphine consumption will record till the postoperative 24 th hours.
  Interventions: Drug: ESP block group
- serratus block group (Active Comparator): Under general anaesthesia, Ultrasound guided SAP block will perform at the T6 level with15 ml bupivacain+ 5ml lidocaine, bilaterally. Morphine 0.1 mg/kg will administer at last 30 minutes of surgery for postoperative analgesia. Patient controlled analgesia (PCA) with morphine will apply to the all patients. Postoperative pain assessment and morphine consumption will record till the postoperative 24 th hours.
  Interventions: Drug: serratus block group

INTERVENTIONS:
Drug: ESP block group — USG guided Erector spinae block (ESP) will perform bilaterally.
  Other Names: USG guided ESP block group
  Arms: ESP block group
Drug: serratus block group — USG guided serratus plane block will perform bilaterally
  Other Names: USG guided serratus plane block
  Arms: serratus block group

SUMMARY:
Total 60 patients, American society of anaesthesiology physical status I-II aged between 18-65 who underwent totally mastectomy will recruit to the study. The patients randomly divided into two groups. Ultrasound guided Erector spinae plane block (ESP) will perform with 15 ml bupivacaine+ 5 ml lidocaine in Group ESP and ultrasound guided serratus anterior plane (SAP) block will perform with 5 ml bupivacaine+ 5 ml lidocaine in Group SAP. Postoperative pain assessment will apply with 11-point numerical rating scale (NRS) and postoperative analgesic requirement will calculate and record with morphine consumption (patient controlled analgesia).

DETAILED DESCRIPTION:
In this study, total 60 patients, American society of anaesthesiology physical status I-II aged between 18-65 who underwent totally mastectomy will recruit. Using with computer randomisation, the patients allocate into two groups. Anaesthesia induction will perform with 2 mg/kg propofol, 0.6 mg/kg rocuronium and 2 microgram/kg fentanil and general anaesthesia will maintain with sevoflurane %1-2 +%40-60 O2-N20 mixture and remifentanil infusion. All of the blocks will perform under general anaesthesia. Ultrasound guided Erector spinae plane block (ESP) will perform with 15 ml bupivacaine+ 5 ml lidocaine in Group ESP and ultrasound guided serratus anterior plane (SAP) block will perform with 5 ml bupivacaine+ 5 ml lidocaine in Group SAP. Postoperative pain, analgesic requirement and complications will evaluate. Postoperative pain assessment will apply with 11-point numerical rating scale (NRS) and postoperative analgesic requirement will calculate and record with morphine consumption (patient controlled analgesia).

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II patients
* Being volunteer
* Total mastectomy

Exclusion Criteria:

* ASA III and over
* Renal and hepatic failure
* Non Volunteers
* Emergency procedures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-09-15 (Estimated); Primary Completion 2019-03-15 (Estimated); Study Completion 2019-04-15 (Estimated)

PRIMARY OUTCOMES:
morphine consumption | up to postoperative 24th hours.
  Patient controlled analgesia (PCA) will provide with morphine PCA. Total morphine consumption will calculate and record till the postoperative 24th hours.

SECONDARY OUTCOMES:
numerical rating scale score | up to postoperative 24th hours.
  Postoperative pain assessment will apply with 11-point numerical rating scale. These scores will record till the postoperative 24 th hours.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Biricik, Principal Investigator — Cukurova University

IPD SHARING:
Plan to Share IPD: No